CLINICAL TRIAL: NCT04918797
Title: A Phase II/III, Open Label, Multicenter Study to Evaluate the Safety, Reactogenicity and Immunogenicity of the Whole-Virion Inactivated SARS-CoV-2 Vaccine (COVAXIN®) in Healthy Volunteers Ages ≤18 to ≥ 2 Years.
Brief Title: COVAXIN in a Pediatric Cohort
Acronym: COVAXIN-Peds
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Bharat Biotech International Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BBIL/BBV152/2021
Record Dates: First submitted 2021-05-18; First posted 2021-06-09 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: SARS-CoV2 Infection
MeSH Terms: conditions — COVID-19 | interventions — BBV152 COVID-19 vaccine

STUDY DESIGN:
Intervention Model Description: Open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study vaccine (Experimental): SARS-COV2 vaccine
  Interventions: Biological: COVAXIN

INTERVENTIONS:
Biological: COVAXIN — Whole-Virion Inactivated SARS-CoV-2 Vaccine (COVAXIN®)

SUMMARY:
The study is designed to evaluate the safety, reactogenicity and immunogenicity of three groups ages ≤18 - >12, ≤12 ->6, ≤ 6 - >2 years of healthy volunteers who receive two doses of the whole virion inactivated SARS-CoV-2 virus vaccine (COVAXIN®) 28 days apart.

Data will be un-blinded to the third party bio-statistician and an interim analysis will be performed on day 56 for Immunogenicity, Safety and submitted to CDSCO.

DETAILED DESCRIPTION:
Study design: A Phase II/III, Open Label, Multicenter Study to Evaluate the Safety, Reactogenicity and Immunogenicity, of the Whole-Virion Inactivated SARS-CoV-2 Vaccine (COVAXIN®) in Healthy Volunteers ages ≤18 to ≥2 Years.

A total sample size of 525 healthy volunteers.

The study is designed to evaluate the safety, reactogenicity and immunogenicity of three groups ages ≤18 - >12, ≤12 ->6, ≤ 6 - >2 years of healthy volunteers who receive two doses of the whole virion inactivated SARS-CoV-2 virus vaccine (COVAXIN®) 28 days apart.

Group1: A total of 175 healthy volunteers ages ≤18->12, years will be enrolled in this group and will receive two doses of BBV152 vaccine through intramuscular route on Day 0 and Day 28+2.

Group 2: A total of 175 healthy volunteers ages ≤12->6, years will be enrolled in this group and will receive two doses of BBV152 vaccine through intramuscular route on Day 0 and Day 28+2.

Group 3: A total of 175 healthy volunteers ages ≤6-> 2 years will be enrolled in this group and will receive two doses of BBV152 vaccine through intramuscular route on Day 0 and Day 28+2.

Data will be un-blinded to the third party bio-statistician and an interim analysis will be performed on day 56 for Immunogenicity, Safety and submitted to CDSCO.

Immunogenicity analysis: A total of 5 ml of blood is collected at days 0, 28+2, 56±7, 118±7 and 208±7. SARS-CoV-2 test will be conducted at the time of screening using RT-PCR and ELISA method.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide written informed consent (by the parents or legally acceptable/authorized representative (LAR) and assent by the children (verbal/oral assent for the children of age between 7-12 years, and written assent for the children of age between >12 to 18 years), and Audio video consent for all participants.
2. Participants of either gender of age between ≥2 to ≤18years (Participant should be ≤18 years at the time of Screening of the study).
3. Good general health as determined by the discretion of investigator.
4. Expressed interest and availability to fulfill the study requirements.
5. Agrees not to participate in another clinical trial at any time during the study period.
6. Agrees to remain in the study area for the entire duration of the study.
7. Willing to allow storage and future use of biological samples for future research.

Exclusion Criteria:

1. History of any other COVID-19 investigational vaccination.
2. Confirmed SARS-CoV-2 at the time of screening using RT-PCR and ELISA method.
3. Temperature >38.0°C (100.4°F) or symptoms of an acute self-limited illness such as an upper respiratory infection or gastroenteritis within three days prior to each dose of vaccine.
4. Receipt of an experimental agent (vaccine, drug, device, etc.) within 60 days before enrollment or expects to receive an investigational agent during the study period.
5. Receipt of any licensed vaccine within four weeks before enrollment in this study.
6. Known sensitivity to any ingredient of the study vaccines, or a more severe allergic reaction and history of allergies in the past.
7. Receipt of immunoglobulin or other blood products within the three months prior to vaccination in this study.
8. Immunosuppression as a result of an underlying illness or treatment with immunosuppressive or cytotoxic drugs, or use of anticancer chemotherapy or radiation therapy within the preceding 36 months.
9. Long-term use (>2 weeks) of oral or parenteral steroids (glucocorticoids) or high-dose inhaled steroids (>800 mcg/day of beclomethasone dipropionate or equivalent) within the preceding six months (nasal and topical steroids are allowed).
10. Any history of hereditary angioedema or idiopathic angioedema.
11. Any history of anaphylaxis in relation to vaccination.
12. History of congenital diseases.
13. Any history of albumin-intolerance.
14. History of any cancer.
15. History of psychiatric severe conditions likely to affect participation in the study.
16. A bleeding disorder (e.g. factor deficiency, coagulopathy or platelet disorder, or prior history of significant bleeding or bruising following IM injections or venepuncture.
17. Any other serious chronic illness requiring hospital specialist supervision.
18. Respiratory diseases like severe acute respiratory syndrome (SARS), including mild asthma.
19. Chronic cardiovascular disease, gastrointestinal disease, liver disease, renal disease, endocrine disorder, and neurological illness
20. History of SARS-CoV-2 infection or known close contact with anyone with laboratory-confirmed SARS-CoV-2 infection or COVID-19 within 2 weeks prior to vaccine administration.
21. Any other condition that in the opinion of the investigator would jeopardize the safety or rights of a volunteer participating in the trial or would render the subject unable to comply with the protocol.

    Re-Vaccination Exclusion Criteria
22. Anaphylactic reaction following administration of the investigational vaccine.
23. Virologically confirmed cases of COVID-19

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 525 (Actual)
Dates: Start 2021-05-26 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2022-01-25 (Actual)

PRIMARY OUTCOMES:
Reactogenicity | Within 7 days after each dose of vaccination
  Occurrence of Solicited Adverse events
Immunogenecity | 6 months
  GMTs of SARS-CoV-2 virus neutralizing antibodies by MNT/PRNT assay.

SECONDARY OUTCOMES:
Immunogenicity | 6 months
  The GMT of binding antibodies (bAb's) IgG against spike protein (S1) and Nucleocapsid (N) protein in all three groups.

OTHER OUTCOMES:
Unsolicited Adverse Events | Within 28 days after each dose of vaccination
  Occurrence of Unsolicited Adverse events
Adverse Events of Special Interest | Through study completion ,an average of 9 months
  Occurrence of Adverse Events of Special Interest

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Vasant Khalatkar, MBBS,MD, Principal Investigator — Meditrina Institute of Medical Sciences,Nagpur; Dr.V.N Tripathi, MBBS,MD, Principal Investigator — Prakhar Hospital Pvt Ltd.,Kanpur; Dr Padmavathi I V, MBBS,MD, Principal Investigator — Victoria Government Hospital; Dr.Lokesh Kumar Tiwari, MBBS,DNB, Principal Investigator — All India Institute of Medical Scienes,Patna; Dr.Jai Prakash Narayan, MBBS,MD, Principal Investigator — JLN Medical college,Ajmer; Dr Mirza Nizam Baig, MBBS,MD, Principal Investigator — Pranam Hospitals Hyderabad; Dr Prashanth Siddiah, MBBS,MD, Principal Investigator — Cheluvambha Hospital,Mysore
Locations (7):
- India (7):
  - Victoria Government Hospital, Visakhapatnam, Andhra Pradesh
  - All India Institute of Medical Sciences, Patna, Bihar
  - Cheluvambha Hospital, Mysore, Karnataka
  - Meditrina Institute of Medical Sciences, Nagpur, Maharashtra
  - Jawahar Lal Nehru Medical college, Ajmer, Rajasthan
  - Pranam Hospitals Hyderabad, Hyderabad, Telangana
  - Prakhar Hospital, Kanpur, Uttar Pradesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vadrevu KM, Reddy S, Jogdand H, Ganneru B, Mirza N, Tripathy VN, Singh C, Khalatkar V, Prasanth S, Rai S, Ella R, Blackwelder W, Prasad S, Ella K. Immunogenicity and reactogenicity of an inactivated SARS-CoV-2 vaccine (BBV152) in children aged 2-18 years: interim data from an open-label, non-randomised, age de-escalation phase 2/3 study. Lancet Infect Dis. 2022 Sep;22(9):1303-1312. doi: 10.1016/S1473-3099(22)00307-3. Epub 2022 Jun 16. PMID 35717995